CLINICAL TRIAL: NCT00500058
Title: A Phase I, Dose-Escalation Study to Assess the Safety and Biological Activity of Recombinant Human Interleukin-18 (SB-485232) Administered by Intravenous Infusion in Combinationwith Rituximab in Adult Patients With B Cell Non-Hodgkin'sLymphoma"
Brief Title: A Phase I, Dose-Escalation Study to Assess the Safety and Biological Activity of Recombinant Human Interleukin-18
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ILI105618
Record Dates: First submitted 2007-07-10; First posted 2007-07-12 (Estimated); Last update posted 2017-07-26 (Actual); Status verified 2017-07

CONDITIONS: Lymphoma, Non-Hodgkin
Keywords: Rituximab,; oncology; IL-18,; combination study,; cytokine,
MeSH Terms: conditions — Lymphoma, Non-Hodgkin; Neoplasms | interventions — Interleukin-18; Rituximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- SB-485232+Rituximab (Experimental): Rituximab 375 milligrams per square meter (mg/m^2) will be administered to subjects with CD20+ B cell lymphoma by intravenous (IV) infusion once a week for four consecutive weeks on Day 1 of Weeks 1 to 4. SB-485232 will be administered by IV infusion over a 2 hour period, at doses ranging from 1 microgram (μg)/kilogram (kg) to 100 μg/kg. SB-485232 will be given once a week for 12 consecutive weeks on Day 2 of Weeks 1 to 4 and Day 2 (± 1 day) of Weeks 5 to 12. SB-485232 will be infused at least 24 hours after the Rituximab infusion was started.
  Interventions: Drug: SB-485232; Drug: Rituximab

INTERVENTIONS:
Drug: SB-485232 — SB-485232 for injection, 7 mg/vial, will be available as a lyophilized cake. It will be reconstituted with 1.4 mL of water for injection. Each vial of this drug product is a clear, colorless solution containing 5 mg/mL of SB-485232.
Drug: Rituximab — Rituximab 375 mg/m^2 will be administered by IV infusion.

SUMMARY:
The purpose is to identify a dose of SB-485232 which is safe, tolerable and effective when used in combination with Rituximab in patients with non-Hodgkin's lymphoma (NHL). This study will use a standard treatment regimen of Rituximab in combination with rising doses of SB-485232. The dose selected from this study will be used in a future studies.

ELIGIBILITY:
Inclusion Criteria:

* Histologically confirmed diagnosis of any subtype of CD20+ B cell NHL. Subjects must have disease that progressed after standard therapy or for which there is no effective standard therapy (including high-dose therapy and autologous stem cell transplantation). NOTE: If the subject has had a prior autologous stem cell transplant, it must have occurred at least three months prior to screening and the subject must be fully recovered from any acute toxicities.
* Prior treatment with Rituximab is allowed, provided it was completed at least six months before study enrollment.
* Male or female ≥ 18 years of age.
* Measurable or evaluable disease.
* Predicted life expectancy of at least 12 weeks.
* ECOG Performance Status of 0 or 1.
* No chemotherapy, immunotherapy, hormonal therapy, or biological therapy for cancer, radiotherapy, or surgical procedures (except for minor surgical procedures) within four weeks before beginning treatment with SB-485232 (6 weeks for nitrosoureas and mitomycin C). Subjects must have recovered from toxicities (incurred as a result of previous therapy) sufficiently to be entered into a Phase I study.
* A signed and dated written informed consent form is obtained from the subject.
* The subject is able to understand and comply with protocol requirements, timetables, instructions and protocol-stated restrictions.

The subject is likely to maintain good venous blood access for PK and PD sampling throughout the study.

* A female is eligible to enter and participate in the study if she is of:

  a. non-childbearing potential (i.e., physiologically incapable of becoming pregnant) including any female who:
* has had a hysterectomy,
* has had a bilateral oophorectomy (ovariectomy),
* has had a bilateral tubal ligation,
* is post-menopausal (demonstrate total cessation of menses for greater than 1year), If amenorrheic for less than one year, post-menopausal status will be confirmed by serum follicle stimulating hormone (FSH) and oestradiol concentrations at screening. or, b. childbearing potential, has a negative serum pregnancy test at the Screen Visit, and agrees to one of the following GSK acceptable contraceptive methods:
* any intrauterine device (IUD) with a documented failure rate of less than

  1% per year.
* vasectomized partner who is sterile prior to the female subject's entry and is the sole sexual partner for that female.
* oral contraceptive (either combined or progesterone only).
* because of the unacceptable failure rate of barrier (chemical and/or physical) methods, the barrier method of contraception must only be used in combination with other acceptable methods described above.
* Adequate organ function,

Exclusion Criteria:

* Women who are pregnant or are breast-feeding.
* Significant cardiac, pulmonary, metabolic, renal, hepatic, gastrointestinal or autoimmune conditions that in the opinion of the investigator and/or GSK medical monitor, places the subject at an unacceptable risk as participant in this trial.
* The subject has diabetes mellitus with poor glycemic control.
* The subject has a history of human immunodeficiency virus (HIV) or other immunodeficiency disease.
* The subject has positive Hepatitis B surface antigen.
* Corrected QT interval (QTc) > 480msec.
* The subject has a history of a severe infusion related reaction or tumor lysis syndrome following treatment with Rituximab (Section 10.2.2).
* The subject has a circulating malignant cell count > 25,000/mm3 in peripheral blood.
* The subject has known anaphylaxis or IgE-mediated hypersensitivity to murine proteins.
* The subject has an acute infection or severe or uncontrolled infections requiring systemic antibiotic therapy.
* Any serious medical or psychiatric disorder that would interfere with subject safety or informed consent.
* Known leptomeningeal disease or evidence of prior or current metastatic brain disease. Routine screening with central nervous system (CNS) imaging studies (CT or MRI) is required only if clinically indicated.
* Receiving concurrent chemotherapy, immunotherapy, radiotherapy, or investigational therapy.
* Oral corticosteroids within 14 days of study entry.
* History of alcohol abuse within six months of screening or alcohol consumption in the past six months exceeding seven drinks/week for women and 14 drinks/week for men (where 1 drink = 5 ounces of wine or 12 ounces of beer or 1.5 ounces of hard liquor).
* History of ventricular arrhythmias requiring drug or device therapy.
* Any unresolved or unstable serious toxicity from prior administration of another investigational drug.
* Any investigational drug within 30 days or five half-lives (whichever is longer) preceding the first dose of SB-485232.
* Donation of blood in excess of 500 mL within a 56-day period prior to dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2007-07-31 (Actual); Primary Completion 2010-03-04 (Actual); Study Completion 2010-03-04 (Actual)

PRIMARY OUTCOMES:
safety/tolerability of combination treatment for 4 weeks safety/tolerability of SB-485232 for additional 8 weeks | 12 weeks

SECONDARY OUTCOMES:
assess blood values of combination treatment for 4 weeks assess blood values of SB-485232 for additional 8 weeks | 12 weeks
Pharmacokinetic parameters for SB-485232 and Rituxan: AUCtau, Cmax, and Cmin. | 12 weeks
Pharmacodynamic biomarker responses: | 12 weeks
Plasma IFN-γ, GMCSF, IP-10, MIG, and MCP-1 changes | from baseline and predose
Plasma IL-18BP change | from baseline
PBMC phenotype changes | from baseline and pre-dose
Activated NK cells (CD16+/CD56+/CD3-/CD69+/FasL+ or IL-18Ra+) | 12 weeks
Activated cytolytic T cells (CD8+/CD4-/CD3+/CD69+ FasL+ or IL- 18Ra+) | 12 weeks
Activated B cells (CD19+/CD25-/CD3-/CD69+) | 12 weeks
Activated Neutrophils/Monocytes (CD11b+/CD16+/CD64+/CD14+/CD45+/CD69+) | 12 weeks
Regulatory T-cells (FoxP3+/CD25+/CD4+/CD127+) | 12 weeks
Immunogenicity (anti-SB-485232 and anti-Rituximab antibodies) | 12 weeks
Anti-tumor activity (Radiographic tumor assessments) | 12 weeks
CD16 (FcγRIIIA) 158V/F genotyping | 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- United States (2):
  - GSK Investigational Site, Chicago, Illinois
  - GSK Investigational Site, Indianapolis, Indiana

IPD SHARING:
Plan to Share IPD: Yes
Patient-level data for this study will be made available through www.clinicalstudydatarequest.com following the timelines and process described on this site.

REFERENCES:
- [Background] Robertson MJ, Kline J, Struemper H, Koch KM, Bauman JW, Gardner OS, Murray SC, Germaschewski F, Weisenbach J, Jonak Z, Toso JF. A dose-escalation study of recombinant human interleukin-18 in combination with rituximab in patients with non-Hodgkin lymphoma. J Immunother. 2013 Jul-Aug;36(6):331-41. doi: 10.1097/CJI.0b013e31829d7e2e. PMID 23799412
- See also: Results for study ILI105618 can be found on the GSK Clinical Study Register. — https://gsk-clinicalstudyregister.com/study/ILI105618?search=study&search_terms=ILI105618#rs
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Study Protocol: ILI105618 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Annotated Case Report Form: ILI105618 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: ILI105618 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Statistical Analysis Plan: ILI105618 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: ILI105618 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: ILI105618 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: ILI105618 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register